CLINICAL TRIAL: NCT03576859
Title: Pyrophosphate Homeostasis and Hepatic Expression of ABCC6. Pilot Study in Liver Transplantation
Brief Title: Pyrophosphate Homeostasis and Hepatic Expression of ABCC6.Pyro-TH
Acronym: Pyro-TH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18-AOI-11
Record Dates: First submitted 2018-06-22; First posted 2018-07-03 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Hepatic Failure
MeSH Terms: conditions — Liver Failure | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cirrhotic patients with chronic liver failure (Other)
  Interventions: Other: blood sample
- cirrhotic patients without chronic liver failure (Other)
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample — Peripheral venous blood is collected before liver transplantation and after restoration of liver function

SUMMARY:
In animals, normal hepatic expression of ABCC6 (ATP-binding transporter cassette, subfamily C, member 6) determines plasma pyrophosphate (PPi) concentration. PPi prevents the formation of hydroxyapatite crystals on tissues by precipitation of calcium and inorganic phosphate (Pi). It is an endogenous compound whose deficiency causes diffuse vascular calcifications in certain rare monogenic diseases, including the elastic pseudoxanthoma caused by the mutation of ABCC6. PPi is produced by enzymatic transformation of extracellular ATP and, in animals, the liver is the main supplier of ATP and PPi (more than 90%). In humans, liver transplantation offers the possibility of correlating the plasma concentration of PPi ([PPi]pl) with hepatic expression of ABCC6. Liver transplantation is performed in the treatment of chronic liver failure (Child B or C) or, in the absence of liver failure, in the treatment of hepatocellular carcinoma. By measuring[PPi]pl before transplantation and after liver function restoration and by measuring ABCC6 in the diseased liver and healthy liver, it is possible to determine whether liver failure is associated with decreased[PPi]pl and decreased liver expression of ABCC6, which is the objective of our pilot study. Its interest is to establish a physiopathological link between the frequent vascular calcifications in obese patients with hepatic steatosis and the production of PPi.

prupose: Look for a deficit in[PPi]pl in patients before the transplant compared to the phase of restoration of liver function

ELIGIBILITY:
Inclusion Criteria:

Indication for liver transplantation Age greater than or equal to 18 years Patients affiliated to social security

Exclusion Criteria:

Patient not affiliated to social security Non-consenting patient or unable to understand the protocol and how it works Fulminant Hepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2020-10-29 (Actual)

PRIMARY OUTCOMES:
plasma PPi concentration between before transplantation and liver function restoration in the both arms | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Untiversity Hospital of Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No